CLINICAL TRIAL: NCT06644482
Title: Exercise as Treatment for Patients With Inclusion Body Myositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Dam Foundation (Other); The Norwegian Rheumatism Association (Other)
Responsible Party: Principal Investigator, Kristine Risum, Senior physioterapist, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 728436
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Inclusion Body Myositis (IBM); Feasibility Study
Keywords: exercise; feasibility study
MeSH Terms: conditions — Myositis, Inclusion Body; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise group in a hospital (Other): Participants will take part in an exercise group delivered once a week in a hospital setting for 16 weeks
  Interventions: Other: Exercise group in a hospital setting

INTERVENTIONS:
Other: Exercise group in a hospital setting — Participants will exercise in a group once a week for 16 weeks in a hospital setting.

SUMMARY:
There is little knowledge about exercise for patients with inclusion body myositis (IBM). Patients with IBM have limited access to rehabilitation and physiotherapy resources, despite a significant need for these services due to the progressive nature of the condition, which leads to a gradual decline in physical function. The purpose of the project is to develop and implement a 16-week exercise intervention at Oslo University Hospital (OUS) for patients with IBM living in Oslo and the surrounding area. The exercise sessions will take place once a week at OUS, under the guidance of physiotherapists with extensive clinical experience with this patient group. Patients are encouraged to exercise at home at least once a week between sessions at OUS to achieve sufficient amount of exercise that normally will improve physical fitness. The feasibility and benefits of the exercise intervention will be evaluated using various methods, such as focus group interviews, physical tests, and questionnaires. The study will also provide valuable insight into whether exercise can lead to improvements in muscle strength, fitness, and balance in patients with IBM.

ELIGIBILITY:
Inclusion Criteria

* IBM diagnosis
* Able to walk with aids

Exclusion Criteria

-Unable to understand and write Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Feasibility: proportion completing the exercise intervention | Baseline to 16 week
  Proportion of included participants completing the exercise intervention
Feasibility: proportion of received exercise diaries | Baseline to 16 weeks
  Proportion of received exercise diaries (0-16 per participant)
Recruitment: proportion enrolled | Baseline
  Proportion of eligible patients enrolled
Feasibility: exercise diaries | Baseline to 16 week
  The participants will log experiences with the intervention (e.g. completed/not completed exercises, reasons for any non-completion, other training activities, barriers/facilitators).
Feasibility: proportion of patients completing physical fitness tests | Baseline and 17 weeks
  Proportion of patients completing physical fitness tests
Feasibilty: Focus group interview | 17 weeks
  Participants will participate in focus group interviews exploring the experiences of the intervention

SECONDARY OUTCOMES:
Changes in walking distance | Baseline and 17 weeks
  Assessed by the 2 minutes walking test. Changes in walking distance measured as meters.
Changes in functional lower extremity strength | Baseline and 17 weeks
  The patients are to stand up and sit down from a chair as many times as they can within 30 seconds, and the total number of times is recorded.
Changes in muscle endurance | Baseline and 17 weeks
  Assessed by the Functional Index- 2 in three muscle groups; shoulder flexors (maximum 60 repetitions), neck flexors (maximum 30 repetitions) and hip flexors (maximum 60 repetitions).
Changes in muscle strength | Baseline and 17 weeks
  Assessed by the Manual Muscle test - 8 (MMT - 8), which includes unilateral testing of muscle strength in 8 eight muscle groups; (Deltoid, Biceps, Wrist extensors, Quadriceps, Ankle dorsiflexors, Neck flexors, Gluteus medius and Gluteus maximux). Each muscle group is scored on a 0-10-point scale (10=best score). The total MMT - 8 will be calculated (0-80, 80=best score).
Changes in grip stength | Baseline and 17 weeks
  Assessed by hydraulic hand dynamometer (Baseline). Change in grip strength is recorded in kilograms.
Change in the Berg Balance Scale | Baseline and 17 weeks
  The Berg Balance Scale (BBS) is a 14-item objective measure that assesses static and dynamic balance and fall risk in adults. Each item is scored on a 5-point ordinal scale ranging from 0 to 4, with 0 indicating an inability to complete the task entirely and 4 indicating an ability to complete the task criterion.The total score ranges from 0-52 (52 indicates best score).
Change in the Inclusion Body Myositis Functional Rating Scale (IBMFRS) | Baseline and 17 weeks
  The IBMFRS consists of 10 questions about a patient's ability to perform daily activities (including walking, dressing, swallowing and handling utensils). Each question is answered using a number from 0-4. The numbers are added up to give the total score ranging from 0 to 40, with 40 being the best possible score
Change in the Health Assessment Questionnaire (HAQ) score | Baseline and 17 weeks
  Change in the last week disability on the total HAQ score (0-3, 0 indicates best possible function). The HAQ comprises 30 questions, covering eight functional ability domains related to daily living during the past week (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities). The score ranges from 0-3 (0 indicates no disability, 3 indicates severe disability) in each domain, of which the total CHAQ is calculated.
Change in Patient Specific Functional Scale (PSFS) | Baseline and 17 weeks
  The patients will identify 3-5 important activities they are unable to perform or have difficulty with due to inclusion body myositis. The patients are then asked to rate the current level of difficulty associated with each activity on an 11-point scale, from 0 (not able to perform the activity) to 10 (no problems).
Change in self-reported physical activity | Baseline and 17 weeks
  Assessed by the International Physical Activity Questionnaire-Short form (IPAQ-SF). Change in time (minutes per week/day) and Metabolic Equivalent of Task (MET-minutes per week/day) spent on sitting, walking, and moderate- and vigorous intensity physical activity the last week. METs are calculated by using the corresponding MET-values for walking (3.3 MET), and moderate-(4.0 MET) and vigorous (8.0 MET) intensity physical activity.
Change in Health-Related Quality of Life | Baseline and 17 weeks
  Assessed by the Short Form Health Survey (SF36) which comprises 36 questions covering the areas of physical function, role limitations (physical), pain, general health perception, energy and fatigue (vitality), social function, role limitations (emotional), and mental health. The results are recoded so that the final score for each area ranges from 0 to 100, where 100 indicates the best possible health.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety]. | Baseline to 16 week
  Patients will log 1) total of falls during the training period and 2) total number of near-falls during the training period.
Incidence of Treatment-Emergent Adverse Events [Tolerability]- pain. | Baseline to 16 week
  Self-reported pain will be assessed by numeric rating scale ranging from 0 (no pain) to 10 (worst pain)
Incidence of Treatment-Emergent Adverse Events [Tolerability]- muscle fatigue | Baseline to 16 week
  Self-reported muscle fatigue will be assessed by numeric rating scale ranging from 0 (no muscle fatigue) to 10 (worst muscle fatigue)
Incidence of Treatment-Emergent Adverse Events [Tolerability]- muscle fatigue | Baseline to 16 week
  Self-reported muscle soreness will be assessed by numeric rating scale ranging from 0 (no muscle soreness) to 10 (worst muscle soreness)
Incidence of Treatment-Emergent Adverse Events [Tolerability]- fatigue | Baseline to 16 week
  Self-reported fatigue will be assessed by numeric rating scale ranging from 0 (no fatigue) to 10 (worst fatigue)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
Data can be made available on reasonable request